CLINICAL TRIAL: NCT05582954
Title: Feasibility and Acceptability of a Guided E-health Programme (EsteemUp), With and Without Gamification Elements, to Increase Self-esteem in University Students.
Brief Title: The Caring Universities Project: EsteemUp RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: VU University of Amsterdam (Other)
Collaborators: Erasmus University Rotterdam (Other); University of Amsterdam (Other); Leiden University (Other); Maastricht University (Other); Utrecht University (Other); InHolland University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Arpana Amarnath, Associate Researcher, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCWE-2022-135
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Self Esteem

STUDY DESIGN:
Intervention Model Description: The present study is a two-armed randomized controlled trial. This trial will be conducted in a university setting. A guided web-based intervention to improve self-esteem (EsteemUp) will be compared to a version of the same intervention with gamification elements (EsteemUp-G)
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent researcher who is not involved in the study will generate the random sequence using a computer random sequence generator. Randomisation will take place at an individual level, stratified by gender and the university where students study. Participants will be randomised into two groups (EsteemUp vs EsteemUp-G) with an allocation ratio of 1:1. We will conduct block randomisation with randomly varied block sizes (6 to 12 allocations per block) to prevent foreknowledge of intervention assignment. Allocation will be concealed from the study's researchers. It is not possible to mask personnel and participants to the treatment allocation because of the nature of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EsteemUp (Experimental): Participants assigned to this arm will receive a 4 week-guided e-health application - EsteemUp - to improve their self-esteem
  Interventions: Behavioral: EsteemUp
- EsteemUp -G (Active Comparator): This group will receive the same intervention (EsteemUp) with the addition of gamification elements.
  Interventions: Behavioral: EsteemUp; Behavioral: EsteemUp-G

INTERVENTIONS:
Behavioral: EsteemUp — EsteemUp is a guided e-health application based on cognitive-behavioural therapy (CBT). It consists of four modules that take approximately 30 to 45 minutes to complete. Each module includes evidence-based psycho-education, reflection questions, interactive exercises, and homework assignments. The content is delivered both textually and visually, including the use of pictures, infographics and videos. Every week trained e-coaches (trained clinical psychology master students) will provide asynchronous written personalized feedback to each participant on the progress of the program and the exercises via the program platform.
Behavioral: EsteemUp-G — The gamification elements added to this arm include (1) Badges - digital rewards upon completing important milestones within the programme EsteemUp. (2) Unlockable content - downloadable worksheets of the exercises that they have done in the module, (3) A certification of completion at the end of the program, (4) Goal setting (5) Gamification terminology - All homework assignments will be framed as a 'challenge' that needs to be completed, (6) a progress bar that will indicate how far along the participant is in the program
  Arms: EsteemUp -G

SUMMARY:
Within the Caring Universities project (study protocol VCWE- 2020-135 accepted by the VCWE), the investigators have developed a guided e-health programme (EsteemUp) designed to increase university students' self-esteem. With the current study, the investigators aim to examine the feasibility and acceptability of EsteemUp - with and without gamification elements - to improve students' self-esteem.

Secondary goals are to gain insight into pre-test to post-test differences regarding self-esteem, symptoms of depression, anxiety and quality of life.

DETAILED DESCRIPTION:
The present study is a two-armed randomized controlled trial. This trial will be conducted in a university setting. Participants will be randomized to receive a version of the intervention either with gamification elements (EsteemUp-G) or without gamification elements (EsteemUp).

EsteemUp was developed based on existing literature on self-esteem and adapted in collaboration with university students to meet the specific needs of the university students. EsteemUp is based on cognitive-behavioural therapy (CBT) and consists of four modules that are delivered via computer, laptop, tablet, or mobile phone. Every module consists of evidence-based information, exercises, and homework assignments. The content is delivered in text format with pictures and infographics. The intervention is available in both English and Dutch.

Participants assigned to EsteemUp-G will receive the exact same intervention explained above with an addition of gamification elements. These elements include Badges, unlockable content, a. certification of completion at the end of the program, goal setting, gamification terminology and a progress bar.

Every week trained e-coaches (trained clinical psychology master students) will provide asynchronous written personalized feedback to each participant on the progress of the program and the exercises via the program platform. Measurements include post-test assessment of adherence, treatment satisfaction, and satisfaction with e-coach. Secondary outcomes include pre and post-assessment of self-esteem, common measures of psychopathology symptoms, and quality of life.

Data will be analysed based on the intent-to-treat principle.

All students currently enrolled at the participating universities (Vrije Universiteit Amsterdam, Erasmus University, InHolland University of Applied sciences, Universities of Amsterdam, Leiden, Utrecht and Maastricht) are potentially eligible for the trial.

Students can participate in EsteemUp free of charge, which will likely increase their self-esteem and confidence. They will not receive any additional incentives for participation.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, a subject must meet all the following criteria:

* Being fluent in Dutch and/or English
* Being enrolled as a student of the seven participating universities
* Being 16 years of age or older
* Having access to a PC or mobile device with internet access
* Provide informed consent before participation

Exclusion Criteria:

- None. All interested students are eligible to participate.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the intervention | T1 (post test: 4-weeks)
  The Client Satisfaction Questionnaire (CSQ-8) is used to measure participants' satisfaction with the overall intervention. The CSQ-8 is commonly used to measure satisfaction with online interventions. It consists of eight items on a four-point Likert scale with a total score ranging from 8 to 32, where a higher score indicates greater satisfaction.
Treatment Adherence | T1 (post test: 4-weeks)
  Adherence refers to "the degree to which the user followed the program as it was designed" (Donkin et al., 2011). The present study measures adherence by dividing the number of modules completed by a participant at time of post-test by the total number of modules in the programme, and multiplying this by 100. The resulting percentage will indicate completion rate.
Satisfaction with E-coach | T1 (post test: 4-weeks)
  The Working Alliance Inventory for guided internet interventions (WAI-I) is used to evaluate participant's satisfaction with the e-coach. The WAI-I consists of 12 items on a 5-point Likert scale with a total score ranging from 12 to 60, where higher scores indicate higher satisfaction

SECONDARY OUTCOMES:
Change in self-esteem | T0 (Baseline) to T1 (Post-test: 4-weeks)
  The Rosenberg Self-Esteem Scale (RSS) is used to measure explicit self-esteem. This tool consists of 10 items measured on a four-point Likert scale ranging from 1(strongly disagree) to 4(strongly agree). The total scores range from 10 to 40 with higher scores indicating better self-esteem.
Change in depressive symptoms | T0 (Baseline) to T1 (Post-test: 4-weeks)
  The Patient Health Questionnaire (PHQ-9) is used as the measure of depression. This questionnaire consists of 9 items scored on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total scores can range from 0 to 27, with higher scores indication more severe depressive symptoms
Change in Anxiety symptoms | T0 (Baseline) to T1 (Post-test: 4-weeks)
  The Generalized Anxiety Disorder scale (GAD-7) is used to measure symptoms of generalized anxiety. The questionnaire consists of 7 items measured on a four-point Likert ranging from 0 (not at all) to 3 (nearly every day). The total scores range from 0 to 21 with higher scores indicating more severe GAD symptoms

OTHER OUTCOMES:
Socio demographic characteristics of participants | T0 (Baseline)
  age gender ethnicity student status study level relationship status whether the student is currently undergoing any treatment (pharmacotherapy/psychotherapy/both/none)
Satisfaction with individual modules | Module 1, Module 2, Module 3, Module 4
  After completing each module, the participants respond to the question "how useful was this module" on a scale of 1 - 100, with higher scores indicating better satisfaction with the module.
Satisfaction with badges | T1 (Post-test: 4-weeks)
  Satisfaction with the badges is measured after completing EsteemUp-G. Participants respond to 3 statements measured on a five-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). These statements are: "The badges were a good addition to the program", "I enjoyed collecting the badges", and "the badges increased my motivation to keep working on the program". The total satisfaction score ranges from 0 to 12, with higher scores indicating greater satisfaction with the badges.

CONTACTS AND LOCATIONS:
Overall Officials: Pim Cuijpers, dr. Prof, Study Director — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands